CLINICAL TRIAL: NCT04692766
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of RPH-104 Treatment in Patients With Idiopathic Recurrent Pericarditis
Brief Title: Study to Evaluate the Efficacy and Safety of RPH-104 Treatment in Patients With Idiopathic Recurrent Pericarditis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Unimed Laboratories (Industry); Data Management 365 (Industry); Center of Pharmaceutical Analytics LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CL04018068
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-104 80 mg (Experimental): subjects will receive RPH-104 at a dose of 80 mg subcutaneously once every 2 weeks
  Interventions: Biological: RPH-104
- Placebo (Placebo Comparator): subjects will receive placebo subcutaneously once every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL transparent glass vial
  Arms: RPH-104 80 mg
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for Injection), 5 mL in a polypropylene ampoule, 10 ampoules per labeled package
  Arms: Placebo

SUMMARY:
The goal of this study was to evaluate the Efficacy and Safety of RPH-104 Treatment in patients in comparison to placebo with Idiopathic Recurrent Pericarditis

DETAILED DESCRIPTION:
The study included the following periods:

1. Screening period (up to 4 weeks); During the screening period, the patients' eligibility for the study was evaluated based on the inclusion/non-inclusion criteria. Those patients who were considered eligible for participation in the study were enrolled in the run-in treatment period.
2. Run-in treatment period (12 weeks, Days 0-84 - for the patients receiving non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine as the therapy for recurrent pericarditis (underlying disease), or 24 weeks, Days 0-168 - for the patients receiving glucocorticosteroids (GCSs) as monotherapy or in combination with NSAIDs and/or colchicine; Depending on the Protocol version, during the period, the patients received the product according to a schedule of 80 mg every two weeks, starting from Day 0 (Protocol version 2.0/3.0). The Protocol amendment (Version 4.0) was accompanied by the adjustment of the treatment regimen and, accordingly, the patients enrolled in the study according to Version 4.0 received the product starting with a loading dose of 160 mg (the first injection on Day 0) and then 80 mg on Day 7, Day 14, and then once every 2 weeks (1 time/2 weeks).

   The treatment response during the run-in treatment period was defined as the resolution of the relapse observed at enrollment in the study, and the absence of new relapses of pericarditis in patients enrolled in the study with signs of pericarditis recurrence; absence of new relapses of pericarditis in patients enrolled without signs of relapse. In the absence of treatment response assessed on Day 14 of the study and then during the preparatory open-label period, the use of RPH-104 in patients was discontinued, and they were prescribed treatment with other drugs at the Investigator's choice.

   After two weeks of open-label therapy (starting from Day 14 of the run-in treatment period), patients with a response to the study drug treatment began to discontinue the previous treatment of the underlying disease. Monotherapy with NSAIDs, colchicine, or their combination was discontinued simultaneously. The GCS dose was gradually tapered over 12 weeks with subsequent complete discontinuation (thus, these patients received RPH-104 in combination with GCS for 14 weeks and RPH-104 as monotherapy for the next 10 weeks).

   The patients who demonstrated response to therapy with RPH-104 during the run-in treatment period, were transferred to the randomized withdrawal period.
3. Randomized withdrawal period (24 weeks: Day 0 since the randomization - Day 168 since the randomization) included treatment with RPH-104 or placebo depending on the randomization group (1:1 ratio) once in 2 weeks and the efficacy and safety monitoring procedures; Patients have been receiving therapy for a period of 24 weeks: the study drug group (to receive RPH-104 80 mg SC) or placebo group (to receive an equivalent volume of placebo subcutaneous (SC)).

   In case of recurrence of pericarditis during the period of randomized withdrawal (regarded as a lack of response), the treatment group was unblinded. Patients in the placebo group were prescribed open-label therapy with RPH-104 as a single dose of 160 mg subcutaneously (first injection), followed by administration of 80 mg every 7 days, 14 days after the first injection. Also, at the Investigator's discretion, the use of NSAIDs and/or colchicine was allowed for relapse treatment in these patients. The response to therapy in such patients was assessed 3 days and 7 days after the first open-label injection of the study drug, according to the results of which, if the relapse was not resolved, the same treatment regimen was continued (including NSAIDs and/or colchicine). Evaluation of the drug efficacy in these patients was carried out 14 days after switching to active study drug treatment. In case of resolution of the developed relapse, the use of NSAIDs/colchicine was to be discontinued simultaneously, the use of the study drug was to be continued at a dose of 80 mg once every other week with an efficacy assessment every 4 weeks until the end of the randomized withdrawal period of the study.

   Patients from the RPH-104 group (as well as patients from the placebo group who were switched to the study drug therapy due to a disease recurrence, those in whom the recurrence did not resolve within 14 days, or patients who developed a new recurrence after the resolution of the previous one) were switched to treatment with other drugs at the discretion of the Investigator; these patients had to come to a follow-up safety visit in 2 and 8 weeks after the administration of the last dose of the study drug.

   Thus, after the end of randomized withdrawal period, the patients who responded to therapy with RPH-104 were asked to transfer to the open-label study to evaluate the long-term safety and efficacy of RPH-104. Non-responders, as well as patients who did not agree to participate in the open-label study of safety and efficacy, had to come to follow-up safety visits.
4. Safety follow-up period included monitoring of safety for 8 weeks after the last dosing of the study drug.

Thus, the maximum duration of treatment in this study was 36 weeks (for patients who were receiving NSAIDs and/or colchicine at the study enrollment) and 48 weeks (as a monotherapy or in combination with NSAIDs and/or colchicine).

The total maximal duration of the study was planned to be approximately 60 weeks.

A total of 20 patients with idiopathic recurrent pericarditis were planned to be randomized into the study. Taking into account potential dropouts during the screening and the run-in treatment period, the number of screened patients (signing the Informed Consent Form) could be as large as 35.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated Informed Consent Form for participation in the study.
* Confirmed diagnosis of idiopathic recurrent pericarditis, established on the basis of the European Society of Cardiology (ESC) diagnostic criteria (2015):

  • The patients may be enrolled in the study with signs of disease recurrence or without them (while on therapy with NSAIDs/GCS/colchicine: any of these drugs or their combinations), but they have to have at least two documented episodes of pericarditis at least 4-6 weeks in between (the second episode can be verified at the moment of the study site visit).
* For patients with signs of relapse, stable therapy (i.e., unchanged dosages and regimen) with NSAIDs/GCSs for not less than 3 days and/or with colchicine for not less than 7 days before screening.
* For patients without signs of relapse: continuous therapy with NSAIDs/GCS/colchicine (any of the drugs or their combination).
* The patient's ability and willingness (in the reasonable opinion of the Investigator) to come to the study site for all scheduled visits, to undergo all study procedures and comply with the protocol requirements, including consent to subcutaneous injections by qualified personnel of the study site.
* Consent of women of childbearing potential (defined as all women with a physiological ability to become pregnant) to use highly effective contraceptive methods throughout the study, starting from the beginning of the screening (signing of the Informed Consent Form) and for at least 8 weeks after discontinuation of the study drug; and the negative pregnancy test result (serum test for chorionic gonadotropin).

OR Consent of sexually active male subjects to use highly effective contraceptive methods throughout the study, starting from the beginning of the screening and for at least 8 weeks after discontinuation of the study drug.

Highly effective methods of contraception include the following:

1. Complete abstinence (if it agrees with the preferable and usual lifestyle of the patient). Periodic abstinence (for example, calendar, ovulation, symptothermal, postovulation methods) and interrupted sexual intercourse are not considered acceptable methods of contraception;
2. Sterilization: surgical bilateral oophorectomy (with or without uterectomy) or ligation of the fallopian tubes at least 6 weeks before the start of the study therapy. If only oophorectomy was performed, the woman's reproductive status should be confirmed by a subsequent assessment of the hormone test;
3. Sterilization of a male partner at least 6 weeks before the start of the study therapy (with proper documented absence of sperm in the ejaculate after vasectomy). In women participating in the study, the sexual partner after vasectomy should be the only partner;
4. use of a combination of any two of the following (a+b or a+c or b+c):

   1. the use of oral, injectable or implanted hormonal contraceptives; in the case of oral contraceptives, women should consistently use the same drug for a minimum of 3 months prior to the initiation of the study treatment;
   2. placement of an intrauterine device (IUD) or intrauterine system (IUS);
   3. barrier methods of contraception: a condom or occlusive cap (diaphragm or cervical/vault caps) and spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

* Hypersensitivity to the study drug (RPH-104), and/or its components/excipients and/or drugs of the same chemical class.
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* Diagnosis of pericarditis of known etiology (tuberculosis-related, tumor-induced, bacterial), rheumatic diseases.
* Other previously diagnosed auto-inflammatory diseases.
* Prior therapy with:
* rilonacept - less than 6 weeks prior to the baseline assessment (Day 0 of the run-in treatment period);
* canakinumab - less than 12 weeks prior to the baseline assessment (Day 0 of the run-in treatment period);
* anakinra - less than 5 weeks prior to the baseline assessment (Day 0 of the run-in treatment period);
* Tumor necrosis factor (TNF) inhibitors, Interleukin 6 (IL-6) inhibitors, Janus kinase inhibitors - less than 12 weeks prior to the baseline assessment (Day 0 of the run-in treatment period);
* immunosuppressive agents (azathioprine, cyclosporine, mycophenolate, mofetil, tacrolimus, sirolimus, mercaptopurine) - less than 24 weeks prior to the baseline assessment (Day 0), methotrexate - less than two weeks prior to the baseline assessment (Day 0),
* any other biological preparations less than 5 half-lives prior to the treatment initiation (Day 0 of the preparatory therapy period).
* The use of live (attenuated) vaccine within 3 months prior to Day 0 (of the run-in treatment period and/or the need to use this type of a vaccine within 3 months after the discontinuation of the study drug. Live attenuated vaccines include vaccines against viral infections such as measles, rubella, mumps, chickenpox, rotavirus, influenza (in the form of a nasal spray), yellow fever, polio (oral polio vaccine); vaccines against tuberculosis (BCG), typhoid (oral typhoid vaccine) and typhus (epidemic typhoid vaccine) vaccines. Patient's immunocompetent family members should refrain from administration of a polio vaccine during the patient's participation in the study.
* Any conditions or signs in the patient that, according to the investigator's judgement, indicate a disorder (suppression) of the patient's immune response and/or significantly increase the risk of immunomodulatory therapy, including, but not limited to, the following:

  * active bacterial, fungal, viral or protozoal infection revealed at the beginning of the screening period;
  * opportunistic infections and/or Kaposi's sarcoma at the beginning of the screening period;
  * chronic bacterial, fungal or viral infection requiring systemic therapy at the beginning of the screening period;
  * HIV-infection, hepatitis B or C (patients with treated hepatitis C and negative polymerase chain reaction (PCR) tests after 3 and 6 months are regarded as cured from hepatitis C and can be included in this study);
  * Disseminated herpes zoster, herpes encephalitis, meningitis, and other non-self-limiting infections caused by the herpes virus within 6 months before the start of the screening period.
* A history of active tuberculosis or the presence of risk factors or signs indicating the presence of active or latent infection caused by M. Tuberculosis, including but not limited to the following:

  * living in specific conditions that increase the risk of contacts with tuberculosis-infected patients, such as prisons, gathering of homeless people etc. over the past year until the beginning of the main treatment period;
  * Occupational exposure at a medical institution in the settings of unprotected contact with patients with a high risk of tuberculosis or patients with tuberculosis during the last year before the start of the screening period;
  * close contact, i.e. being in the same room (at home or in another confined environment) for an extended period of time (days or weeks rather than minutes or hours) with a person with active pulmonary tuberculosis within the past year prior to the beginning of the treatment period;
  * test results indicating active tuberculosis or latent infection caused by M. Tuberculosis: positive result of QuantiFERON-TB/T-SPOT test.TB during the screening period; findings of chest X-ray exam in two views confirming pulmonary tuberculosis during the screening period.
* The presence of any other significant comorbidities (cardiovascular, nervous, endocrine, urinary tract, gastrointestinal tract, liver, blood clotting disorders, other autoimmune diseases, etc.) or conditions that may, in the reasonable opinion of the Investigator, adversely affect the participation and well-being of the study subject and/or distort the evaluation of the study results.
* History of organ transplantation or the need for transplantation surgery at the beginning of the screening period, or elective transplant surgery during the study.
* Any malignant neoplasms during the screening period or within 5 years before its onset, except for non-metastatic basal cell and squamous cell carcinoma after complete resection or carcinoma in situ of any type after complete resection.
* Mental disorders that, in the reasonable opinion of the Investigator, may affect the patient's participation in the study or his/her ability to comply with the Protocol procedures.
* Pregnancy or breast-feeding
* History of abuse of alcohol or psychoactive substances as assessed by the Investigator.
* Severe renal impairment: creatinine clearance by Cockcroft-Gault formula <30 mL/min at the screening.
* Concomitant participation in other clinical studies at the moment of the beginning of the screening or the use of any not approved (investigational) medicinal products within 4 weeks of 5 half-life periods (depending on what is longer) up to the baseline assessment (Day 0 of the run-in treatment period).
* Presence of any of the following at the screening:
* Absolute neutrophil count <1.5 х 10^9/L,
* white blood cells (WBC) count <3.5 х 10^9/L,
* platelet count <100 х 10^9/L,
* hemoglobin ≤ 80 g/L,
* glycated hemoglobin (HbA1c) ≥ 8% (to be evaluated only in patients with diabetes mellitus),
* alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 3.0 х upper limit of normal (ULN),
* Total bilirubin >1.5 х ULN (except for cases of documented Gilbert's syndrome)
* Previous participation in this clinical study, provided that at least one dose of the study drug was administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Time (days) to the recurrence within 24 weeks after randomization | up to 24 weeks after randomization
  Time (days) to the recurrence within 24 weeks after randomization in patients with idiopathic recurrent pericarditis treated with RPH-104 compared to placebo.

SECONDARY OUTCOMES:
Proportion of patients demonstrating a response to RPH-104 treatment | Day 3, Day 7, Day 14 of the run-in treatment period
  Proportion of patients demonstrating a response to RPH-104 treatment on Day 3, Day 7, Day 14 of the run-in treatment period
The proportion of patients switched to active treatment with RPH-104 | Day 3, Day 7, Day 14 of the run-in treatment period
  The proportion of patients switched to active treatment with RPH-104 due to the development of a relapse during the period of randomized withdrawal, with a response to treatment in 3 days, 7 and 14 days after the study drug administration.
Proportion of patients with pericarditis recurrence throughout the run-in treatment period | up to 24 weeks
  Proportion of patients with pericarditis recurrence throughout the run-in treatment period.
Proportion of patients, treated with RPH-104 with pericarditis recurrence recurrence within 24 weeks after the randomization, compared to placebo. | up to 24 weeks
  Proportion of patients, treated with RPH-104, with pericarditis recurrence within 24 weeks after the randomization, compared to placebo.
Proportion of patients who completely discontinued corticosteroids within 12 weeks following the response to therapy throughout the run-in treatment period. | up to 24 weeks
  Proportion of patients who completely discontinued corticosteroids within 12 weeks following the response to therapy throughout the run-in treatment period
Change in chest pain from baseline assessed by the patients during the run-in treatment period | from Day 0 up to 24 weeks
  Change in chest pain from baseline (Day 0 of the run-in treatment period) assessed by the patients using a numeric rating scale (NRS) during the run-in treatment period.
  NRS contains 11 values from 0 to 10 points, where 0 is no pain, 10 is unbearable pain.
Change in chest pain assessed by the patients during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change in chest pain from the assessment on the Day 0 of the randomized withdrawal period assessed by the patients using NRS during the randomized withdrawal period in patients treated with RPH-104 compared to placebo.
  NRS contains 11 values from 0 to 10 points, where 0 is no pain, 10 is unbearable pain.
Change in C-reactive protein (CRP) level during the run-in treatment period | from Day 0 of up to 24 weeks
  Change in C-reactive protein (CRP) level from baseline (Day 0 of the run-in treatment period) during the run-in treatment period.
Change in C-reactive protein (CRP) level during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change of the CRP level from Day 0 of the randomized withdrawal period during the randomized withdrawal period for RPH-104 administration versus placebo.
Change of the size of pericardial effusion from baseline based on echocardiography (Echo-CG) data during the run-in treatment period | from Day 0 up to 24 weeks
  Change of the size of pericardial effusion from baseline (Day 0 of the run-in treatment period) based on Echo-CG data during the run-in treatment period.
Change of the size of pericardial effusion from baseline based on Echo-CG data during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change of the size of pericardial effusion according to the echocardiography data from Day 0 of the randomized withdrawal period during the randomized withdrawal period for RPH-104 administration versus placebo.
Change in physician global assessment of disease activity from baseline assessed using a numeric rating scale during the run-in treatment period | from Day 0 up to 24 weeks
  Change in physician global assessment of disease activity from baseline (Day 0 of the run-in treatment period) assessed using a numeric rating scale during the run-in treatment period.
  Global disease activity is assessed by the physician using a NRS containing 11 values from 0 to 10 points, where 0 is the absence of active disease, 10 is the maximum activity of the disease.
Change in physician global assessment of disease activity assessed using a numeric rating scale during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change in physician global assessment of disease activity from the assessment on the Day 0 of the randomized withdrawal period assessed using a numeric rating scale during the randomized withdrawal period in patients treated with RPH-104 compared to placebo.
  Global disease activity is assessed by the physician using a NRS containing 11 values from 0 to 10 points, where 0 is the absence of active disease, 10 is the maximum activity of the disease.
Change in patient's overall health self-assessment during the run-in treatment period | from Day 0 up to 24 weeks
  Change from baseline (Day 0 of the preparatory therapy period) of the patient's overall health self-assessment on the numerical rating scale during the preparatory therapy period.
  The patient's overall health is assessed using a NRS containing 11 values from 0 to 10 points, where 0 is very good, 10 is very poor.
Change in patient's overall health self-assessment during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change of the patient's overall health self-assessment on the numerical rating scale from Day 0 of the randomized withdrawal period during the randomized withdrawal period of RPH-104 administration versus placebo.
Change in quality of life from baseline based on data of the SF-36 questionnaire during the run-in treatment period | from Day 0 up to 24 weeks
  Change in quality of life from baseline (Day 0 of the run-in treatment period) based on data of the SF-36® questionnaire during the run-in treatment period
Change in quality of life based on data of the SF-36 questionnaire during the randomized withdrawal period | from Day 0 of the randomized withdrawal period up to 24 weeks
  Change in quality of life from the assessment on the Day 0 of the randomized withdrawal period based on data of the SF-36 questionnaire during the randomized withdrawal period in patients treated with RPH-104 compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (2):
- Russia (2):
  - Federal Budgetary Healthcare Institution Orenburg Regional Clinical Hospital, Orenburg
  - Federal State Budget Institution "V.A. Almazov National Medical Research Center" of Ministry of Healthcare of Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myachikova VY, Maslyanskiy AL, Moiseeva OM, Vinogradova OV, Gleykina EV, Lavrovsky Y, Abbate A, Grishin SA, Egorova AN, Schedrova ML, Samsonov MY. Treatment of Idiopathic Recurrent Pericarditis With Goflikicept: Phase II/III Study Results. J Am Coll Cardiol. 2023 Jul 4;82(1):30-40. doi: 10.1016/j.jacc.2023.04.046. PMID 37380301